CLINICAL TRIAL: NCT03912805
Title: Clinical Trial to Evaluate ET-01 in Subjects With Lateral Canthal Lines
Brief Title: ET-01 in Subjects With Lateral Canthal Lines, LCL-209
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-01-LCL-209
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Lateral Canthal Lines, LCL; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: vehicle controlled, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle, topical liniment, administered once at baseline
  Interventions: Biological: Vehicle
- ET-01 1610U (Experimental): botulinum toxin, Type A, topical liniment, administered once at baseline
  Interventions: Biological: botulinum toxin, Type A

INTERVENTIONS:
Biological: botulinum toxin, Type A — topical liniment
  Other Names: ET-01 1610U
  Arms: ET-01 1610U
Biological: Vehicle — Vehicle Formulation
  Arms: Vehicle

SUMMARY:
This study tests an investigational drug formulation called ET-01, botulinum toxin, Type A, topical, in lateral canthal lines (LCL).

DETAILED DESCRIPTION:
This product is being tested for its ability to reduce lateral canthal lines (LCL), also known as Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* females 25 - 65 years of age
* minimal to moderate Crow's Feet wrinkles at rest
* moderate to severe Crow's Feet on contraction
* adequate vision to assess facial wrinkles in a mirror
* willingness to refrain from products affecting skin remodeling
* female subjects must be not pregnant and non-lactating
* subjects should be in good general health

Exclusion Criteria:

* history of adverse reactions to any prior botulinum toxin treatments
* history of vaccination or non-response to any prior botulinum toxin treatments
* botulinum toxin treatment in the prior 6 months
* present or history of neuromuscular disease, eyelid ptosis, muscle weakness, paralysis, or "dry eye"
* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Synexis, Inc., Pinellas Park, Florida
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three medical centers between February 2019 and October 2019
Pre-assignment Details: A total of N=45 subjects were screened; N=38 were found eligible; N=7 subjects screen failed prior to treatment assignment; N=38 were randomized
Groups:
- ET-01 1610U: botulinum toxin, Type A, topical liniment, administered once at baseline
  botulinum toxin, Type A: topical liniment, 1610U
Period: Overall Study
Arm/Group | Vehicle | ET-01 1610U
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | ET-01 1610U | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 38
IGA-C [Mean (Standard Deviation); unit: units on a scale] — Investigator Global Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.4 (0.5) | 3.4 (0.5) | 3.4 (0.5)
SSA-C [Mean (Standard Deviation); unit: units on a scale] — Subject Self-Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.6 (0.5) | 3.5 (0.5) | 3.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response Defined as Change in IGA-C (Investigators Global Assessment) Score by at Least 2 Ordinals From Baseline to Week 4
Description: Investigators Global Assessment of the Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe). Response is defined as change by at least two ordinals from Baseline to Week 4.
Time Frame: Week 4
Population: Intent-To-Treat (ITT) population defined as all treated subjects who reached Week 4. No imputation was performed when only incomplete data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | ET-01 1610U
Number analyzed (Participants) | 19 | 19
Participants | 3 | 1

2. Secondary Outcome: Total Number of Observations With a Response Defined as Change ≥2 in IGA-C and SSA-C Score at Any Post Baseline Visit
Description: Total number of observations with a change in the Investigators Global Assessment on Contraction, IGA-C, and the Subject Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as a change by at least two ordinals in both assessments. The observation period includes all post-baseline visits from Week 1 to Week 26.
Time Frame: Week 1, 2, 4, 8,12,18, and 26
Population: Total number of observations with a change in the Investigators Global Assessment on Contraction, IGA-C, and the Subject Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as a change by at least two ordinals in both assessments. The observation period includes all post-baseline visits from Week 1 to Week 26.
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | ET-01 1610U
Number analyzed (Participants) | 19 | 19
Number analyzed (Observations) | 132 | 132
Observations | 8 | 12

3. Secondary Outcome: Total Number of Observations With a Response Defined as Change in SSA-C Score ≥ 2 at Any Post Baseline Visit
Description: Total number of observations with a change in the Subject Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as a change by at least two ordinals in both assessments. The observation period includes all post-baseline visits from Week 1 to Week 26.
Time Frame: Week 1, 2, 4, 8,12,18, and 26
Population: Intent-To-Treat (ITT) population defined as all treated subjects who had at least one post-baseline visit. No imputation was performed when only incomplete data were available.
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | ET-01 1610U
Number analyzed (Participants) | 19 | 19
Number analyzed (Observations) | 132 | 132
Observations | 15 | 20

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Vehicle | ET-01 1610U
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 6/19 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=19) | ET-01 1610U (N=19)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thermal Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Endodontic Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Oral Herpes (General disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Results are considered Confidential Information that may not be published or disclosed without Sponsor's written consent for a period of five (5) years after completion of the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03912805/Prot_SAP_000.pdf